CLINICAL TRIAL: NCT05083962
Title: Healthy Lifestyle Program: A Novel Group-based Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Richard J. Joseph, M.D., MD, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002707
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Lifestyle Program Intervention Arm (Active Comparator)
  Interventions: Behavioral: Healthy Lifestyle Program
- Waitlist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Healthy Lifestyle Program — An intensive behavior change curriculum designed to help create and sustain healthy habits
  Arms: Healthy Lifestyle Program Intervention Arm

SUMMARY:
The Healthy Lifestyle Program involves twelve, 2-hour seminars during which participants will learn how to build healthy behaviors through a combination of individual and group exercises. Participants will use lessons from the seminars to pursue health goals and learn the basics of physical fitness, nutrition, sleep & recovery, stress management, and weight management for optimal health. Throughout the program, participants will be supported by a behavior coach along with dedicated fitness training, dietary strategy, and stress management support. As part of this next installment of the program, we are conducting a study of the Healthy Lifestyle Program to capture outcome data, including weight/BMI, blood pressure, hemoglobin A1c, and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Preferential access to the HLP is provided folks who live in the neighborhoods of Roxbury, Dorchester, and Mattapan. However, this is certainly not exclusive and we continue to have participants from all around the greater Boston area, especially now that the program is being delivered virtually.

Exclusion Criteria:

* There are no groups of people who are excluded from participating in the program, except for the specified by the age cut offs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
BMI | 1 year

IPD SHARING:
Plan to Share IPD: No